CLINICAL TRIAL: NCT01598454
Title: Phase 1 Study on the Use of Racotumomab Anti-idiotype Antibody in Patients With Pediatric Malignancies That Express N-glycolylated Gangliosides and Are Resistant to Conventional Treatment.
Brief Title: Use of Racotumomab in Patients With Pediatric Tumors Expressing N-glycolylated Gangliosides
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR-RACO-1-2-09
Record Dates: First submitted 2012-05-10; First posted 2012-05-15 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Neuroblastoma; Ewing's Sarcoma; Wilm's Tumor; Retinoblastoma; Glioma
MeSH Terms: conditions — Neuroblastoma; Sarcoma, Ewing; Wilms Tumor; Retinoblastoma; Glioma | interventions — racotumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Racotumomab (Experimental)
  Interventions: Drug: racotumomab

INTERVENTIONS:
Drug: racotumomab — Dosage form: intradermal injection. Dosage: 0.15 mg; 0.25 mg; 0.4 mg. Frequency: 3 biweekly injections or 6 biweekly injections. Duration: 4 weeks or 10 weeks.

SUMMARY:
This study will be carried out in children with diagnosis of cancer with tumors known to express N-glycolylated gangliosides. The disease must be resistant to conventional therapy. The acute toxicity and immune response will be evaluated.

The expression of N-glycolylated gangliosides in tumors has previously been investigated in the tumor sample bank at this Hospital. The expression of N-glycolyl GM3 was shown in neuroblastoma, Ewing's sarcoma, Wilm's tumor and retinoblastoma.

Gliomas and the aforementioned tumor types have a very bad prognosis when conventional treatment is ineffective.

New therapeutic strategies have thus been examined, and several immunotherapeutic approaches, including dendritic cell vaccines, peptide vaccines and anti-idiotype vaccines are currently being assessed.

Racotumomab is an anti-idiotype antibody capable of inducing anti-N-glycolyl GM3 antibodies in patients with melanoma, breast cancer and lung cancer.

Dose escalation studies have shown the safety of racotumomab in the 0.5 to 2 mg dose range. The 1 mg dose level was selected for the ensuing clinical studies.

This clinical trial in children involves three dose levels: 0.15 mg, 0.25 mg and 0.4 mg, owing to the difference in body surface between an adult (1.73 sq. m in average) and the candidate population for this study (0.55 to 0.7 sq. m).

ELIGIBILITY:
Inclusion Criteria:

* Children (both genders) of between 1 and 10 years old at the time of accrual.
* Diagnosis of neuroblastoma (progression after first line treatment), glioma (progressing disease or metastatic disease, without curative treatment options), Ewing's sarcoma (progressive metastatic disease to first line treatment or progressive disease to second line treatment), Wilm's tumor (metastatic relapse after treatment), or retinoblastoma (progressing disease or metastatic relapse during or after first line treatment).
* Previous cancer treatment finished 30 days before accrual.
* Lansky performance status over 50.

Exclusion Criteria:

* History of encephalopathy, convulsions, asthma or severe allergy.
* Infectious disease grade 3 or 4 according to CTCAE version 3.
* Hepatic, kidney or cardiac insufficiency.
* Marrow insufficiency after self-transplantation of hematopoietic stem cells.
* Weight inferior to 12 kg at the time of accrual.
* Concomitant cancer treatment.
* Inability to comply with study procedures.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2011-02; Primary Completion 2014-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Selection of the higher safe dose level for ensuing clinical trials | Up to 1 year
  One of the three dose levels assessed in this study will be selected for further clinical testing in children: 0.15 mg, 0,25 mg or 0.4 mg.

SECONDARY OUTCOMES:
Assess the immune response to racotumomab treatment | Up to 1 year
  Active specific immunotherapy with racotumomab has shown to elicit antigen-specific immune responses in adult patients. The elicitation of anti-immunogen and anti-ganglioside antibodies will be assessed in serum samples prior and after racotumomab treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Cacciavillano, MD, Principal Investigator — Prof. Dr. J. P. Garrahan National Children's Hospital; Guillermo Chantada, MD, Study Director — Prof. Dr. J. P. Garrahan National Children's Hospital
Locations (1):
- Prof. Dr. J. P. Garrahan National Children's Hospital, Buenos Aires, Argentina

REFERENCES:
- [Result] Cacciavillano W, Sampor C, Venier C, Gabri MR, de Davila MT, Galluzzo ML, Guthmann MD, Fainboim L, Alonso DF, Chantada GL. A Phase I Study of the Anti-Idiotype Vaccine Racotumomab in Neuroblastoma and Other Pediatric Refractory Malignancies. Pediatr Blood Cancer. 2015 Dec;62(12):2120-4. doi: 10.1002/pbc.25631. Epub 2015 Jul 7. PMID 26154941
- See also: Prof. Dr. J. P. Garrahan National Children's Hospital — http://www.garrahan.gov.ar